CLINICAL TRIAL: NCT04735185
Title: Randomized, Comparative-effectiveness Study of Intradiscal Autologous Bone Marrow Concentrate Versus Intradiscal Corticosteroid for Chronic Discogenic Low Back Pain
Brief Title: Stem Cells vs. Steroids for Discogenic Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in protocol per FDA that required funding and logistics that could not be accommodated.
Sponsor: Johns Hopkins University (Other)
Collaborators: The Geneva Foundation (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00250806
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Chronic Low Back Pain; Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Adrenal Cortex Hormones; Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: We are trying to determine whether intradiscal injection of autologous BMC (bone marrow-derived mesenchymal stem cells) will decrease pain and improve function compared with intradiscal steroid.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradiscal autologous stem cells (Active Comparator): Participants in this arm will have autologous stem cells harvested through bone marrow aspiration. The stem cells that were harvested will be processed and injected into affected intradiscal spaces in the lumber spine.
  Interventions: Other: Autologous stem cells
- Intradiscal corticosteroid and local anesthetic (Active Comparator): Participants in this arm will receive an intradiscal injection of the steroid methylprednisolone and the local anesthetic bupivacaine into affected intradiscal spaces in the lumber spine.
  Interventions: Drug: Corticosteroid; Drug: Local anesthetic

INTERVENTIONS:
Other: Autologous stem cells — In this intervention participants will receive a 2 mL intradiscal injection into each affected disc of autologous bone marrow-derived mesenchymal stem cells from bone marrow aspirate of the posterior ilium.
  Arms: Intradiscal autologous stem cells
Drug: Corticosteroid — In this intervention participants will receive a 1 mL intradiscal injection of the steroid methylprednisolone (40 mg/mL) into each affected disc.
  Arms: Intradiscal corticosteroid and local anesthetic
Drug: Local anesthetic — In this intervention participants will receive a 1 mL intradiscal injection of the local anesthetic bupivacaine 0.5% into each affected disc.
  Arms: Intradiscal corticosteroid and local anesthetic

SUMMARY:
This is a randomized, comparative-effectiveness study comparing intradiscal autologous stem cells (from bone marrow aspirate) to intradiscal corticosteroid for the treatment of chronic discogenic low back pain (LBP). The primary objective of this study is to determine whether intradiscal autologous stem cells (from bone marrow aspirate) is more effective than intradiscal steroids for the treatment of chronic discogenic low back pain (LBP). Participants in this study will be randomized to receive up to intradiscal stem cell injections at 1 or 2 discs with cells harvested from a bone marrow aspirate drawn from participants' iliac crest, or an equal volume (2 mL) of intradiscal steroids and local anesthetic injected into the discs. In order to identify the painful disc(s), discography may be used at the discretion of the provider. Both treatments are frequently used as part of clinical care (i.e. there is no placebo group).

DETAILED DESCRIPTION:
In this study, the investigators are attempting to determine if intradiscal injection of autologous bone marrow-derived mesenchymal stem cells (BMC) will decrease pain and improve function compared with intradiscal steroids.

Up to 106 patients with a clinical diagnosis of chronic discogenic low back pain for greater than 6 months, MRI evidence of lumbar disc degeneration limited to one or two discs with <50% disc height loss, and positive provocative discography (if clinically indicated) will be randomized to receive intradiscal BMC or steroid and long-acting local anesthetic (bupivacaine).

Those randomized to group I will receive a 2 mL intradiscal injection of autologous bone marrow-derived mesenchymal stem cells from bone marrow aspirate of the posterior ilium, while those randomized to group II will receive an intradiscal injection of the steroid methylprednisolone and the local anesthetic bupivacaine. The first follow-up will occur at 4-weeks post-treatment at which time rescue medications may be prescribed or adjusted but no other analgesic interventions should occur. The primary outcome measure will be pain relief at 3 months post-treatment, while a positive categorical outcome will be a 2-point or greater decrease in average LBP coupled with either a score > 5/7 on the PGIC (indicating noticeable improvement) or a 10-point decrease in ODI (indicating a clinically meaningful benefit). At 3 months, a repeat MRI will be obtained in selected patients at military treatment facilities (i.e. every 5th patient). Those who fail to experience a positive categorical outcome will be withdrawn from the study to receive alternate care, including an option for intradiscal BMC in those who received corticosteroid. For those who continue to experience a positive outcome, there will be 6- and 12-month follow up visits. At all follow-up visits, histories and physical exams will be performed and questionnaires assessing sleep, function, and anxiety and depression will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Pain duration > 6 months
3. Failure of non-operative treatment > 3 months
4. Average pain score > 4/10 over the past week
5. Presumed clinical diagnosis of discogenic low back pain (such as back>leg pain, no or minimal radiation of pain past knee level, no significant improvement with epidural steroid injection, facet injections, sacroiliac joint injections and/or trigger point injections
6. Lumbar MRI within the last 18 months showing disc degeneration in <= 2 lumbar discs; <50% disc height loss in each disc
7. Patient agrees to have disc injection(s) and no other low back interventional or pharmacological treatments for at least 3 months
8. Patient agrees to be off all NSAIDs and corticosteroids from 2 weeks prior to and 3 months after the injection.
9. Stable dose of analgesic medications for at least 2 weeks

Exclusion Criteria:

1. Previous disc directed therapy involving heat (e.g. Intradiscal electrothermal therapy (IDET), biacuplasty)
2. Previous disc injection therapy in the last 3 months (e.g. corticosteroid, platelet rich plasma, stem cells)
3. Previous lumbar spine surgery (e.g. discectomy, fusion) at the affected levels (i.e. those with relief after surgery in whom adjacent segment discogenic pain is suspected can be considered on a case-by-case basis)
4. Disc extrusion or symptomatic disc protrusion at affected level
5. Untreated coagulopathy
6. Allergy to contrast dye or local anesthetics
7. Negative discography or discography showing > 2 positive discs
8. Pain > 15 years in duration
9. Opioid dose > 30 mg oral morphine equivalents per day (patients may be tapered down or off opioids)
10. Diffuse pain phenotype (e.g. diagnosis of fibromyalgia)
11. Secondary gain (e.g. ongoing medical board or litigation related to injury)
12. Pregnancy (study subject report of negative pregnancy status will be sufficient to participate. Testing will be provided if subject is unsure or requests a test to confirm.
13. Cannot read or understand English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in average low back pain score on 0-10 numerical rating scale | Baseline and 3 months
  Mean change in average low back pain score over the past week at 3 months compared to baseline on 0-10 numerical rating scale (higher pain scores represent greater pain)

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale score | 4 weeks
  14-question scale measuring anxiety and depression, with each question scored as 0-3 (higher numbers represent greater anxiety or depression).
Hospital Anxiety and Depression Scale score | 3 months
  14-question scale measuring anxiety and depression, with each question scored as 0-3 (higher numbers represent greater anxiety or depression).
Hospital Anxiety and Depression Scale score | 6 months
  14-question scale measuring anxiety and depression, with each question scored as 0-3 (higher numbers represent greater anxiety or depression).
Hospital Anxiety and Depression Scale score | 1 year
  14-question scale measuring anxiety and depression, with each question scored as 0-3 (higher numbers represent greater anxiety or depression).
Athens Insomnia Scale score | 4 weeks
  Scale measuring sleep dysfunction on an 8-question 0-24 scale, with higher numbers indicating greater dysfunction.
Athens Insomnia Scale score | 3 months
  Scale measuring sleep dysfunction on an 8-question 0-24 scale, with higher numbers indicating greater dysfunction.
Athens Insomnia Scale score | 6 months
  Scale measuring sleep dysfunction on an 8-question 0-24 scale, with higher numbers indicating greater dysfunction.
Athens Insomnia Scale score | 1 year
  Scale measuring sleep dysfunction on an 8-question 0-24 scale, with higher numbers indicating greater dysfunction.
Patient global impression of change (PGIC) score | 4 weeks
  1-7 scale evaluating, with higher scores indicating greater improvement.
Patient global impression of change (PGIC) score | 3 months
  1-7 scale evaluating, with higher scores indicating greater improvement.
Patient global impression of change (PGIC) score | 6 months
  1-7 scale evaluating, with higher scores indicating greater improvement.
Patient global impression of change (PGIC) score | 1 year
  1-7 scale evaluating, with higher scores indicating greater improvement.
Oswestry disability index score | 4 weeks
  0-100% score measuring function for back and/ leg pain (higher scores indicate worse function)
Oswestry disability index score | 3 months
  0-100% score measuring function for back and/ leg pain (higher scores indicate worse function)
Oswestry disability index score | 6 months
  0-100% score measuring function for back and/ leg pain (higher scores indicate worse function)
Oswestry disability index score | 1 year
  0-100% score measuring function for back and/ leg pain (higher scores indicate worse function)
Disc Degeneration based on MRI | 3 months
  Disc degeneration on MRI (graded as significantly improved, slightly improved, no change, and worsening degeneration, based on Pfirmann's scale).
Average low back pain score on 0-10 numerical rating scale | 4 weeks
  Average low back pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain).
Average low back pain score on 0-10 numerical rating scale | 3 months
  Average low back pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain).
Average low back pain score on 0-10 numerical rating scale | 6 months
  Average low back pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain).
Average low back pain score on 0-10 numerical rating scale | 1 year
  Average low back pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain).
Mean change in worst low back pain score on 0-10 numerical rating scale | Baseline and 4 weeks
  Mean change in worst low back pain score over the past week at week 4 compared to baseline on 0-10 numerical rating scale (higher pain scores represent greater pain).
Mean change in worst low back pain score on 0-10 numerical rating scale | Baseline and 3 months
  Mean change in worst low back pain score over the past week at week 3 months compared to baseline on 0-10 numerical rating scale (higher pain scores represent greater pain).
Mean change in worst low back pain score on 0-10 numerical rating scale | Baseline and 6 months
  Mean change in worst low back pain score over the past week at week 6 months compared to baseline on 0-10 numerical rating scale (higher pain scores represent greater pain).
Mean change in worst low back pain score on 0-10 numerical rating scale | Baseline and 1 year
  Mean change in worst low back pain score over the past week at week 1 year compared to baseline on 0-10 numerical rating scale (higher pain scores represent greater pain).
Worst low back pain score on 0-10 numerical rating scale | 4 weeks
  Worst low back pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain).
Worst low back pain score on 0-10 numerical rating scale | 3 months
  Worst low back pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain).
Worst low back pain score on 0-10 numerical rating scale | 6 months
  Worst low back pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain).
Worst low back pain score on 0-10 numerical rating scale | 12 months
  Worst low back pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain).
Positive categorical outcome | 4 weeks
  Greater or equal to 2-point decrease in average low back pain score coupled with a PGIC score of 5 or higher or a decrease on Oswestry disability score of 10 or greater
Positive categorical outcome | 3 months
  Greater or equal to 2-point decrease in average low back pain score coupled with a PGIC score of 5 or higher or a decrease on Oswestry disability score of 10 or greater
Positive categorical outcome | 6 months
  Greater or equal to 2-point decrease in average low back pain score coupled with a PGIC score of 5 or higher or a decrease on Oswestry disability score of 10 or greater
Positive categorical outcome | 12 months
  Greater or equal to 2-point decrease in average low back pain score coupled with a PGIC score of 5 or higher or a decrease on Oswestry disability score of 10 or greater

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be available upon request per approval of the U.S. Department of Defense (DoD).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: For up to 3 years
Access Criteria: Per approval by the funding organization (U.S. Department of Defense)

REFERENCES:
- [Background] Pettine KA, Murphy MB, Suzuki RK, Sand TT. Percutaneous injection of autologous bone marrow concentrate cells significantly reduces lumbar discogenic pain through 12 months. Stem Cells. 2015 Jan;33(1):146-56. doi: 10.1002/stem.1845. PMID 25187512
- [Background] Noriega DC, Ardura F, Hernandez-Ramajo R, Martin-Ferrero MA, Sanchez-Lite I, Toribio B, Alberca M, Garcia V, Moraleda JM, Sanchez A, Garcia-Sancho J. Intervertebral Disc Repair by Allogeneic Mesenchymal Bone Marrow Cells: A Randomized Controlled Trial. Transplantation. 2017 Aug;101(8):1945-1951. doi: 10.1097/TP.0000000000001484. PMID 27661661